CLINICAL TRIAL: NCT04443842
Title: Effectiveness of Behavioural Economics-based Incentives on Glycaemic Control and Lifestyle in Adults With Newly Diagnosed Type 2 Diabetes: a Feasibility Pilot Study
Brief Title: Behavioural Economics-based Incentives in Adults With Type 2 Diabetes Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BET2-v2-202005
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive the usual standard care (same as control group), loss-framed financial incentive, social incentives and weekly feedback on performance for 6 months.
  Interventions: Behavioral: Financial and social incentives
- Control (No Intervention): Participants will receive standard care including patient screening and education on diet, physical activity, and smoking conducted by a multi-disciplinary team. Participants in the control group will neither be told their baseline step count nor receive any feedback messages.

INTERVENTIONS:
Behavioral: Financial and social incentives — Participants will be credited with HK$1000 in their virtual accounts at the beginning of the trial. After baseline step counts are gathered in the second week, participants will lose HK$40 for each subsequent week that they do not meet their personal weekly step target.
  The social incentives are peer comparison and social support. Participants receive feedback of their physical activity performance by assessing whether they met or exceeded their step count target, followed by positive messages for encouragement. Nominated supporters will be informed of participants' performance for social support.
  Arms: Intervention

SUMMARY:
A feasibility pilot study of a randomised control trial of adults newly diagnosed with type 2 diabetes to compare the effectiveness of financial and social incentives on healthy lifestyle behaviour.

DETAILED DESCRIPTION:
This is a pilot study of testing the feasibility of the interventions being implemented in our main trial in local settings. Adults newly diagnosed with type 2 diabetes without receiving any anti-diabetic medication in Hong Kong are randomised to compare the effectiveness of financial and social incentives against a control group receiving standard care. The investigators follow participants for 9-months (6-month intervention period and a 3-month post-intervention follow-up period) to assess glycemic control and other health indicators. Participants will be randomly assigned to one of two groups (in ratio 3:1): arm A (financial and social incentives in addition to standard care), and arm B (control arm receiving standard care). Financial incentives will be framed around loss aversion and the endowment effect. Social incentives will include peer competition, and social support. Financial and social incentives are to encourage increased physical activity and participants will use a pedometer to track activity. Participants are followed for an additional 3-months after the cessation of incentives to assess the sustainability of lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adults aged 30-70 years
* Capable of providing informed consent
* Resident in Hong Kong
* Able to communicate in English or Chinese
* Newly diagnosed with type 2 diabetes within a year according to World Health Organization guidelines: HbA1c ≥ 48 mmol/mol (≥ 6.5%); fasting plasma glucose ≥ 7.0 mmol/l (≥ 126 mg/dl); oral glucose tolerance test (OGTT) ≥ 11.1 mmol/l (200 mg/dl) with symptoms, or on two separate occasions if asymptomatic
* HbA1c ≤ 7.5%
* Not taking any medication for glycaemic control
* Willing to take blood tests
* Access to a smart phone to track physical activity
* Physically mobile for duration of the trial

Exclusion Criteria:

* Already participating in another intervention study
* Any health condition prohibiting them from completing the 9-month trial, such as history of eating disorder, cancer, serious illness, breastfeeding
* Medical conditions that can affect HbA1c measurements including anaemia, haemoglobinopathies, haemodialysis, iron/B12 deficiency or supplements, chronic liver diseases, splenectomy, rheumatoid arthritis, use of anti-retroviral drugs, ribavirin, or aspirin
* Intend to receive medication for glycaemic control in the next 6 months
* Intend to seek private medical treatment for diabetes in the next 6 months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Baseline, 6 and 9 months
  Change in HbA1c levels

SECONDARY OUTCOMES:
Change in physical activity (step count) | Baseline, 6 and 9 months
  Step counts
Change in body weight | Baseline, 6 and 9 months
  kg
Changes in lipid profile | Baseline, 6 and 9 months
  Total, HDL- and LDL-cholesterol; Triglycerides
Change in physical activity level | Baseline, 6 and 9 months
  International Physical Activity Questionnaires (IPAQ)

OTHER OUTCOMES:
Change in health service utilisation | Baseline, 6 and 9 months
  Number of attendances and hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Jianchao Quan, MPH, BM BCh, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- School of Public Health, Li Ka Shing Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Information will shared in accordance with the University of Hong Kong Data Management Plan (DMP)
Supporting Information: Study Protocol, SAP
URL: https://hub.hku.hk/researchdata/staff2.htm